CLINICAL TRIAL: NCT01169623
Title: Assessing The Effect Of Educational Intervention Based On Supportive Behaviour Leadership Model On Head Nurses' Performance In TUMS Hospitals: RCT In 2010
Brief Title: Effect Of Educational Intervention Based On Supportive Leadership
Acronym: EEIBSL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mandana Shirazi, Assistant Professor of Tehran University of Medical Science, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10292 TUMS
Record Dates: First submitted 2010-07-14; First posted 2010-07-26 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2010-01

CONDITIONS: The Effects of Educational Intervention on Nurses Performance
Keywords: Supportive leadership behaviour; Nurse Performance; Educational Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Intervention (Experimental): 55 of head nurses who will participate in educational Intervention arm based on supportive leadership behaviour model
  Interventions: Other: Assessing the Effect Of Educational Intervention Based On Supportive Leadership Behavior on Iranian head nurses leadership performance
- CONTROL (Placebo Comparator): 55 of head nurses who will not participate in educational intervention will be considered as a control arm
  Interventions: Other: Assessing the Effect Of Educational Intervention Based On Supportive Leadership Behavior on Iranian head nurses leadership performance

INTERVENTIONS:
Other: Assessing the Effect Of Educational Intervention Based On Supportive Leadership Behavior on Iranian head nurses leadership performance — 55 of head nurses who will participate in educational Intervention arm based on supportive leadership behaviour model

SUMMARY:
Hypothesis Applying Educational Intervention Based On Supportive behaviour Leadership Model has positive effect on Head Nurses' performance in TUMS Hospitals.

Specific objectives

1. Assessing the impact of supportive leadership behaviour on individual head nurse
2. Assessing the impact of supportive leadership behaviour on nursing team
3. Assessing the impact of supportive leadership behaviour on TUMS organizational success, especially in cross-functional environments
4. Develop a specific plan for effectively supportive leadership behaviour the efforts of others to sustain and encourage productive performance and employee satisfaction

DETAILED DESCRIPTION:
Methods Design and Setting In this randomized controlled intervention study, the participants of intervention group attended a one day multifaceted supportive leadership workshop, designed for head nurses, working in academic hospitals of Tehran University of Medical Sciences (TUMS).

Supportive leadership behaviors were assessed, by the use of a new developed and validated instrument. The subordinates' points of view were assessed in both control and intervention groups before the intervention and three months after it. Head and subordinate nurses from the sixteen main metropolitan academic hospitals of TUMS were included. This study was performed from July 2010 to April 2011. (Figure1).

Participants A number of 110 head nurses were selected by the use of stratified randomized sampling among 235 head nurses in 16 metropolitan academic hospitals. Moreover, six subordinates were considered for each head nurse (660 subordinates) with different levels of nursing education such as Registered Nurse and Nurse Aids. Therefore, the total number of participants was 770. The sampling processes were conducted with the help of 16 nurse managers (matrons) in these 16 hospitals. Individuals were included into the study based on inclusion criteria. In order to avoid bias, these 16 nurse managers were excluded from the study population (Figure 2). The response rate was 95% in baseline phase as a result of face to face visit. The inclusion criteria was for nurses having more than two month work experience in the same ward and the intention of staying in that position for an additional three month.

The head nurses and their related subordinates (660 subordinates) were randomized into an intervention and a control group. The researchers were blinded during randomization. The head nurses in the intervention group (n=55) participated in a multifaceted course of supportive leadership style, and the head nurses in the control group (n=55) did not receive any training. All 770 participants were blinded about their group and completed the questionnaires in baseline and after the intervention. Up to 39 subordinate participants were excluded from the study due to a change in their hospital work place; and the rest of the participants (n= 731) filled out the questionnaires in the post -test. The variables consisted of supportive leadership behavior (SLB), age, sex, marital status and employment background.

Ethical statement This study was approved by the University Ethical Committee and registered as a clinical trial in Clinical Trial.gov (NCT 01169623) and all the participants in the study signed the informed consent. .

Intervention Intervention was performed based on a multifaceted learning and teaching style in the intervention group. The intervention consisted of a one day eight hour workshop held at the Educational Development Center (EDC) of TUMS, twice with 25 to 27 head nurses participating in each workshop. The contents and expected outcomes of the workshop were emerged from the concepts of different leadership styles, including fundamentals of supportive leadership behavior, and some parts of a similar workshop held in Canada (Toronto University (2008) entitled:" Practical Approach To Giving Recognition").

To increase the effectiveness of the workshops, we used an interactive multifaceted approach. The teaching methods included role playing, mini-lectures, and modified gold fish bowl. First, the workshop began with the ice breaking method introducing workshop's participants and facilitatorsto each other. Then, a 30 minute mini lecture was presented regarding current terminology of leadership and its' difference with managing by an expert in the field. Following that, the participants were encouraged to discuss about the "subject., Then the session continued with a 15 minute lecture regarding different types of leadership (task oriented leader, behaviorist leader,…) and their strengths and weaknesses. During the workshop, we had conducted three role playing relay on three different scenarios based on different leadership styles and managerial dilemma in hospitals performed by our simulated nurse managers and nursing staffs. . They were carried out through the goldfish bowl technique, known as a small group technique in medical education. This method had previously been used in changing behaviors such as communication skills, problem solving through creative and indirect approach and alternative approaches to practice dilemma (Mohanna et al., 2003, p 81; Thistlethwaite & Ridgway, 2006, p 23), Then participants discussed the role playing, reflected on the actors' roles and talked about their points of view. Also, participants were expected to distinguish between different leadership behaviors and styles and select one based on the workshop program. Finally the facilitators of the workshop summarized the discussions and gave the participants a feedback regarding each role playing and focused on the important learning objectives based on the leadership style. The workshop targeted to introduce supportive leadership in comparison with other leadership styles and its strong points.

Questionnaires The main instrument in this study was the SLB questionnaire. Since there was no valid and reliable instrument to assess specifically SLB, and none of them were adapted or developed in nursing context, the provisional questions of this instrument were extracted by experts from SLB questions of three different questionnaires: Ohio State (OSQ) (Larsson 2006), Developmental Leadership (DL) (Hersey & Blanchard 1979), and Hersey and Blanchard's Situational theory (HBS) (Halpin 1962) are three valid and common generic scales related to leadership styles. Some of their items which were related to SLB were extracted from these questionnaires. Those items were translated into Farsi and also back translated to English by two separate bilingual English language experts. Moreover, some new questions were developed and added to the first draft, which led to a 50-item questionnaire in total. The content and face validity of the instrument was ensured through discussion and consensus within the group of experts. The reliability of the questionnaire was assessed using a test-retest approach in pilot study, conducted among 30 of nurses, and then they were excluded from main population. Kappa coefficient were used for assessing the correlation between test and retest results. All the items with Kappa less than 0.7 were excluded from the final version. The second version of questionnaire was comprised of forty items, and the mean Kappa for all questionnaires was 0.86. The internal consistency of SLB scale as measured by Cronbach's alpha was 0.84. The second version of instrument,comprised of 40 items in four dimension of supportive leadership: support for development (18 items of 40-item questionnaire), integrity (a 7 item subscale that reflect trustworthiness, encouragement and good interpersonal communication skill), sincerity (8 items which showed high quality loading on demonstrating friendly and approachable behaviors) and recognition (a 7 item subscale that asked about supportive environment which everyone is recognized and appreciated). An exploratory factor analysis was conducted based on principle axis factoring and Varimax rotation to evaluate the construct validity of scale. The Cronbach's alpha for each factors were above 0.3(range 0.3-0.9).

ELIGIBILITY:
1. Working in the ward more than 2 months
2. To work at university hospital depend to Tehran University of Medical Sciences
3. Asking and be assuring about continuing their job at least for next three month
4. Asking their age, gender, work experience

Exclusion criteria

1. do not want to cooperate in this project
2. some nurses who intend to move to another places after 2 month
3. nurses who were not ready to filling out the the questionnaires due to their movement to another ward

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Supportive leadership behaviour questionnaire for assessing head nurses performance | 10 months
  110 head nurses of TUMS performance will be assessed through their subordinates, who were answering to the questionnaire. we have considered 6 subordinates for each head nurse. The total number of assessment will be 660 before and 660 after interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Shirazi, PhD, Study Chair — University Tehran
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Shirazi M, Emami AH, Mirmoosavi SJ, Alavinia SM, Zamanian H, Fathollahbeigi F, Masiello I. The effects of intervention based on supportive leadership behaviour on Iranian nursing leadership performance: a randomized controlled trial. J Nurs Manag. 2016 Apr;24(3):400-8. doi: 10.1111/jonm.12335. Epub 2015 Sep 29. PMID 26416084